CLINICAL TRIAL: NCT07350655
Title: Effect of Virtual Reality-based Training on Postural Stability in Patients With Chronic Non-specific Low Back Pain
Brief Title: Efficacy of Virtual Reality-based Training in Patients With Chronic Non-specific Low Back Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Hosam Magdy Metwally, Assistant professor of physical therapy, Al-Ahliyya Amman University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 100099
Record Dates: First submitted 2025-12-23; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Non Specific Chronic Low Back Pain
Keywords: virtual reality-based training; postural stability; chronic non-specific low back pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality-based training (Other): Group A receives virtual reality-based training and assessment using the Biodex Balance System and the forward reach test
  Interventions: Device: VR (VR-Control)
- balance exercises (Other): Group B receives balance exercises and assessment using the Biodex Balance System and the forward reach test
  Interventions: Other: Balance training

INTERVENTIONS:
Device: VR (VR-Control) — uses immersive, computer-generated environments and virtual reality headsets to simulate real-world situations, allowing trainees to practice skills in a safe, interactive, and risk-free setting. This technology offers advantages like cost savings, reduced risk in hazardous situations, better learning retention through hands-on experience, and the ability to repeat scenarios for proficiency.
  Arms: virtual reality-based training
Other: Balance training — Balance exercises that can help with low back pain include single-leg standing, heel-to-toe walking, calf raises, bird-dogs, and bridges, which strengthen the core muscles and improve overall stability. Start by holding onto a sturdy object for support and gradually increase the difficulty by moving to less stable surfaces or closing your eyes.
  Arms: balance exercises

SUMMARY:
Low back pain is one of the most prevalent pain conditions worldwide. Virtual reality-based training has been explored as a new treatment strategy for low back pain. Present evidence indicates that the effectiveness of virtual reality-based training for people with chronic low back pain is inconclusive.

All patients will be recruited from the faculty of physical therapy at the October 6 University All the assessment measurements will be done at the Faculty of Physical Therapy, October 6 University

ELIGIBILITY:
Inclusion Criteria:

1. All patients will suffer from mechanical low back pain
2. Age will range from 30 to 40 years 3 - All patients will have a BMI range of 25-29

Exclusion Criteria:

1. History of radicular pain
2. Lumbar discs prolapse.
3. Visual problems
4. History of previous lumbar surgery
5. BMI more than 29

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Biodex balance system | one week
  The Biodex Balance System (BBS) has been used to evaluate postural balance. The BBS is a multiaxial device that objectively measures and records an individual's ability to stabilise the involved joint under dynamic stress. It uses a circular platform that is free to move in the anterior-posterior and medial-lateral axes simultaneously
Forward reach test | one week
  The forward reach test is a clinical assessment that measures a person's ability to reach forward while standing in a fixed position to gauge their stability and fall risk. To perform the test, a patient stands next to a wall with their arm raised and fist closed, and they reach as far as possible along a yardstick or meter stick without moving their feet or losing their balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Ahliyya Amman University, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No